CLINICAL TRIAL: NCT07140900
Title: A Phase 1b Open-label, Multicenter Study Evaluating the Safety, Tolerability, and Efficacy of Xaluritamig in Combination With Androgen Receptor Pathway Inhibitors in Participants With Metastatic Hormone-sensitive Prostate Cancer
Brief Title: Study Evaluating the Safety, Tolerability, and Efficacy of Xaluritamig in Combination With Androgen Receptor Pathway Inhibitors in Participants With Metastatic Hormone-sensitive Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240361
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Keywords: Prostate cancer; Xaluritamig
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xaluritamig with Darolutamide (Experimental): Participants will receive xaluritamig in combination with darolutamide. Participants will enter long-term follow-up for up to 3 years from the first dose of study treatment, or until withdrawal of consent, lost to follow-up, or participant death, whichever occurs first.
  Interventions: Drug: Xaluritamig; Drug: Darolutamide
- Xaluritamig with Abiraterone (Experimental): Participants will receive xaluritamig in combination with abiraterone. Participants will enter long-term follow-up for up to 3 years from the first dose of study treatment, or until withdrawal of consent, lost to follow-up, or participant death, whichever occurs first.
  Interventions: Drug: Xaluritamig; Drug: Abiraterone

INTERVENTIONS:
Drug: Xaluritamig — Participants will receive xaluritamig intravenously.
  Other Names: AMG 509
Drug: Darolutamide — Participants will receive darolutamide orally.
  Arms: Xaluritamig with Darolutamide
Drug: Abiraterone — Participants will receive abiraterone orally.
  Arms: Xaluritamig with Abiraterone

SUMMARY:
The main objective of the trial is to evaluate the safety and tolerability of xaluritamig in combination with darolutamide or abiraterone.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate. Mixed histologies (eg, adenocarcinoma with neuroendocrine component) are not permitted.
* Participants must have at the time of diagnosis:

  * De novo mHSPC, defined as metastatic disease with no prior diagnosis of localized prostate cancer AND started androgen deprivation therapy (ADT) (luteinising hormone-releasing hormone [LHRH] agonist/antagonist or orchiectomy) with or without androgen receptor pathway inhibitor (ARPI) (defined as abiraterone OR darolutamide) as SOC, first treatment with ADT should be no longer than 12 weeks before screening. Prior docetaxel treatment is not permitted.
* Participants must have at the time of diagnosis:

  * High-volume metastatic disease defined as presence of visceral metastasis and/or ≥ 4 bone metastases with at least one outside of the vertebral column and pelvis.
* Documented metastatic disease either by a positive bone scan, or for soft tissue or visceral metastases, either by contrast enhanced abdominal/pelvic/chest computed tomography (CT) or magnetic resonance imaging (MRI) scan.
* PSA not progressing per PCWG3 following the initial PSA nadir after starting ADT.

Exclusion Criteria:

* Prior history of central nervous system (CNS) metastases.
* Unresolved toxicities from prior anti-tumor therapy (excluding those related to ongoing ADT and ARPI) not having resolved to Common Terminology Criteria for Adverse events (CTCAE) version 5.0 grade 1 or baseline, with the exception of alopecia or toxicities that are stable and well-controlled AND there is an agreement to allow inclusion by both the investigator and the sponsor.
* Autoimmune disease requiring systemic immunosuppression within the past 2 years.
* Participant with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active or systemic infection within 7 days prior to the first dose of study treatment.
* Prior six-transmembrane epithelial antigen of the prostate 1 (STEAP1)-targeted therapy.
* Prior radioligand therapy (RLT), poly-adenosine diphosphate ribose polymerase (PARP) inhibitor, cytotoxic chemotherapy, aminoglutethimide or ketoconazole for prostate cancer, or any prior systemic biologic therapy, including immunotherapy for prostate cancer.
* Prior enzalutamide or apalutamide within 15 days prior to enrollment.
* Requirement for chronic systemic corticosteroid therapy (prednisone dose greater than 10 mg per day or local equivalent) or any other immunosuppressive therapies (including anti TNFα therapies) unless stopped (with adequate tapering) within 7 days prior to dosing.
* Prior radiotherapy (to the prostate and/or to all visible metastatic lesions in a metastasis-directed therapy approach); palliative radiation within 2 weeks prior to first dose of study treatment is allowed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-04-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | Up to approximately 2.5 years
Number of Participants with Treatment-related Adverse Events | Up to approximately 2.5 years
Number of Participants with Clinically Significant Changes in Vital Signs | Up to approximately 2.5 years
Number of Participants with Clinically Significant Changes in Clinical Laboratory Tests | Up to approximately 2.5 years

SECONDARY OUTCOMES:
Percentage of Participants with Prostate-specific Antigen (PSA) < 0.2 ng/mL at 6 Months | 6 months
Time to PSA Progression | Up to approximately 4.5 years
Time to First New Systemic Anticancer Therapy | Up to approximately 4.5 years
Time to Radiographic Progression per Prostate Cancer Working Group 3 (PCWG3) Modified Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to approximately 4.5 years
Observed Concentration at the End of a Dose Interval of Darolutamide | Up to approximately 4.5 years
Observed Concentration at the End of a Dose Interval of Abiraterone | Up to approximately 4.5 years
Maximum Observed Serum Concentration (Cmax) of Xaluritmag | Up to approximately 4.5 years
Time to Cmax (Tmax) of Xaluritmag | Up to approximately 4.5 years
Area Under the Concentration Time Curve (AUC) of Xaluritmag | Up to approximately 4.5 years
Half-life (t1/2) of Xaluritamig | Up to approximately 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
- Australia (5):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Cabrini Hospital, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Switzerland (3):
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Sankt Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this trial will be considered beginning 18 months after the trial has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this trial.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen trial/trials in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com